CLINICAL TRIAL: NCT01758601
Title: Estudio de intervención Nutricional Para la evaluación de Los Beneficios Sobre la Salud Derivados Del Consumo de Merluza en población Con Alto Riesgo Cardiovascular.
Brief Title: White Fish for Cardiovascular Risk Factors in Patients With Metabolic Syndrome: the WISH-CARE Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Collaborators: CIBER de Fisiopatología de la Obesidad y Nutrición (CIBERobn). (Unknown); Pescanova S.A., Pontevedra, Spain. (Unknown)
Responsible Party: Principal Investigator, Jose I. Botella-Carretero, MD, PhD, MBA, Clinical Assistance, Clinical Researcher, MD, PhD., Hospital Universitario Ramon y Cajal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: WISH-CARE
Record Dates: First submitted 2012-12-27; First posted 2013-01-01 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Cardiovascular Risk Factors; Metabolic Syndrome
Keywords: white fish; Metabolic syndrome; Cardiovascular risk
MeSH Terms: conditions — Metabolic Syndrome | interventions — Diet Therapy; Seafood

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fish - no fish (Experimental): The individuals randomized to this arm continued with their previous alimentary habits, avoiding any significant nutritional imbalance, and with an ingestion of 7 serves of hake (each serve consisted of 100g of frozen Namibia hake, Pescanova S.A., Pontevedra, Spain) per week for a period of 8 weeks. Then switched to previous alimentary habits, avoiding any significant nutritional imbalance, as well as any fish or seafood.
  Interventions: Other: Dietary intervention with 7 servings oh white fish per week (each serve consisted of 100g of frozen Namibia hake, Pescanova S.A., Pontevedra, Spain); Other: Previous alimentary habits, avoiding any significant nutritional imbalance, as well as any fish or seafood
- No fish - fish (Active Comparator): Patients were on previous diet except for the avoidance of fish and any other seafood for 8 weeks. Afterwards they were changed to the same diet but with 7 serves of hake per week.
  Interventions: Other: Dietary intervention with 7 servings oh white fish per week (each serve consisted of 100g of frozen Namibia hake, Pescanova S.A., Pontevedra, Spain); Other: Previous alimentary habits, avoiding any significant nutritional imbalance, as well as any fish or seafood

INTERVENTIONS:
Other: Dietary intervention with 7 servings oh white fish per week (each serve consisted of 100g of frozen Namibia hake, Pescanova S.A., Pontevedra, Spain)
Other: Previous alimentary habits, avoiding any significant nutritional imbalance, as well as any fish or seafood

SUMMARY:
The investigators performed this study to evaluate the efficacy of regular ingestion of white fish to reduce cardiovascular risk factors in patients with the metabolic syndrome, compared to a diet with no fish or seafood at all.

DETAILED DESCRIPTION:
This study was designed as a randomized cross-over multicenter clinical trial with participating centers from the CIBER de Fisiopatología de la Obesidad y Nutrición (CIBERobn), coordinated by the Hospital Universitario Ramón y Cajal, Madrid. The investigators included adult patients with the metabolic syndrome as defined by the Third Report of the National Cholesterol Education Program, Adult Treatment Panel III. All the subjects were Caucasian from European ancestry. Patients were randomized after the screening visit to one of two sequences: 1) Sequence 1 to receive fish consumption first and then no fish. The individuals randomized to this arm continued with their previous alimentary habits, avoiding any significant nutritional imbalance, and with an ingestion of 7 serves of hake (each serve consisted of 100g of frozen Namibia hake, Pescanova S.A., Pontevedra, Spain) per week for a period of 8 weeks. Afterwards they continued for another 8 weeks with the same diet except for the avoidance of fish and any other seafood; 2) Sequence 2 for which they started with their previous alimentary habits, avoiding any significant nutritional imbalance, as well as any fish or seafood for the first 8 weeks. Afterwards they were changed to the same diet but with 7 serves of hake per week.

ELIGIBILITY:
Inclusion Criteria:

* We included adult patients with the metabolic syndrome as defined by the Third Report of the National Cholesterol Education Program, Adult Treatment Panel III.

Exclusion Criteria:

* Fish allergy and positive antibodies to Anisakis spp.
* Morbid obesity with BMI ≥40kg/m2.
* Chronic renal failure.
* Chronic psychopathy.
* Neoplasia.
* Refusal to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Serum lipids | 8 WEEKS
  The primary outcome was to study the effects of hake consumption on lipid profiles, particularly on serum triglycerides.

SECONDARY OUTCOMES:
Other individual components of the metabolic syndrome, C-reactive protein, fatty acids, insulin-resistance. | 8 weeks
  The secondary outcomes were: the benefits on the other individual components of the metabolic syndrome, apart from lipids, as defined by the ATPIII (waist circumference, blood pressure levels, and glycemia); the effects on serum pro-inflammatory markers such as C-reactive protein, and also on insulin-resistance as calculated by the homeostasis model assessment; to identify specific biomarkers of white-fish consumption associated with the encountered benefits in patients with metabolic syndrome, specifically by measuring serum fatty acids.

OTHER OUTCOMES:
Omega-3 fatty acids in random subgroup. | 8 weeks
  To identify specific biomarkers of white-fish consumption associated with the encountered benefits in patients with metabolic syndrome, specifically by measuring serum fatty acids.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Vazquez C, Botella-Carretero JI, Corella D, Fiol M, Lage M, Lurbe E, Richart C, Fernandez-Real JM, Fuentes F, Ordonez A, de Cos AI, Salas-Salvado J, Burguera B, Estruch R, Ros E, Pastor O, Casanueva FF; WISH-CARE Study Investigators. White fish reduces cardiovascular risk factors in patients with metabolic syndrome: the WISH-CARE study, a multicenter randomized clinical trial. Nutr Metab Cardiovasc Dis. 2014 Mar;24(3):328-35. doi: 10.1016/j.numecd.2013.09.018. Epub 2013 Nov 1. PMID 24462043